CLINICAL TRIAL: NCT04051593
Title: Cervical Stabilization Exercises Improved Pain, Disability, and Physical Impairments in University Violinists With Nonspecific Neck Pain
Brief Title: Effects of Cervical Stabilization Exercise in Violinists With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, YI-JU TSAI, Associate Professor, National Cheng Kung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NationalCheng-KungU
Record Dates: First submitted 2019-08-03; First posted 2019-08-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain
Keywords: cervical stabilization exercise
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Exercise
  Interventions: Other: Cervical stabilization exercise

INTERVENTIONS:
Other: Cervical stabilization exercise — The participants followed instructional videos and performed the cervical stabilization exercise program at home for 20 minutes/day, 3 days/week, for 6 weeks.

SUMMARY:
The purpose of this study is to examine the influence of a 6-week cervical stabilization exercise program in university violin players with chronic nonspecific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* duration of playing the instrument longer than 5 years
* practicing the violin more than 5 hours/week
* constant neck pain for more than 3 months or at least 2 pain episodes in the last 3 months

Exclusion Criteria:

* previous surgery in the neck and shoulder regions
* current participation in a structured exercises program
* current treatment for neck and shoulder pain
* red flags suggesting of cancer, infection, vascular insufficiency, and etc. during history taking
* neurological symptoms of the upper extremities during screening tests (e.g. Spurling test and upper limb tension tests)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported neck pain: Numeric Rating Scale | Pre-test 1 (week 0), Pre-test 2 (week 4) and Post-test (week 10)
  Measured by the Numeric Rating Scale (min 0-max 10, better outcome 0 worst outcome 10)
Changes in neck disability | Pre-test 1 (week 0), Pre-test 2 (week 4) and Post-test (week 10)
  Measured by the Neck Disability Index (10-item questionnaire, each item scored from 0 to 5, result expressed as percentage, better outcome 0 worst outcome 100%)

SECONDARY OUTCOMES:
Changes in deep neck flexors function | Pre-test 1 (week 0), Pre-test 2 (week 4) and Post-test (week 10)
  Measured by the craniocervical flexion test with a pressure biofeedback unit (higher pressure represents better outcome)
Changes in cervical muscle endurance | Pre-test 1 (week 0), Pre-test 2 (week 4) and Post-test (week 10)
  Measured using a stopwatch for the successful time holding the head in cervical flexion and extension positions (longer time represent better outcome)
Changes in cervical joint position sense | Pre-test 1 (week 0), Pre-test 2 (week 4) and Post-test (week 10)
  Measured by the cervcal joint reposition error with a laser pointer (short distance represent better outcome)
Changes in upper body posture | Pre-test 1 (week 0), Pre-test 2 (week 4) and Post-test (week 10)
  Evaluated by the photographic method

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ju Tsai, Ph.D., Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04051593/Prot_SAP_000.pdf